CLINICAL TRIAL: NCT04395066
Title: Molecular Diagnosis and Prognosis of Severe Pulmonary Infection in Immunosuppressed Hosts
Brief Title: Molecular Diagnosis and Prognosis of Severe Pulmonary Infection Immunosuppressed Hosts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ruilan Wang, PhD, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 2018KY149
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Severe Pneumonia; Immunosuppressed Hosts; Diagnosis
MeSH Terms: conditions — Pneumonia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CD55 — CD55 is an important complement regulatory protein that inhibits C3 and C5 activation by blocking the formation and accelerating the decay of new C3 and C5 convertases, both of which mediate downstream actions of all three complement activation pathways, and CD55 protects host cells from complement attack.

SUMMARY:
Serious pneumonia is a serious inflammation of the lungs caused by various pathogens, resulting in severe bacteraemia or toxemia, which in turn causes blood pressure drop, shock, blurred consciousness, restlessness, delirium and coma, etc., and requires intensive care and treatment in intensive care unit (ICU) because of its seriousness. There is an upward trend in the number of clinically immunosuppressed host patients, including long-term use of glucocorticoids for rheumatoid immune diseases and kidney diseases, tumor chemotherapy, organ transplantation, etc. A huge risk for these patients is the diagnosis and treatment of infections, especially lung infections. We have previously observed a significant increase in mortality from severe pneumonia in immunosuppressed patients, and our recent analysis of 204 patients with novel coronavirus pneumonia found that low lymphatic counts, immunosuppression, etc. were independent risk factors for death in patients. Early diagnosis and timely treatment are the main means to reduce the mortality rate of severe pneumonia. CD55 is an important complement regulatory protein that inhibits C3 and C5 activation by blocking the formation and accelerating the decay of new C3 and C5 convertases, both of which mediate the downstream action of all three complement activation pathways, and CD55 protects host cells from complement attack. Our previous study found that CD55 was significantly elevated in patients with severe pneumonia. Therefore, this project proposes "Early diagnosis of severe pneumonia based on combination of biomarkers with new generation pathogenesis and early clinical manifestations". It is proposed to validate the predictive effects of recently discovered markers such as CD55, HBP and CD64 on severe pneumonia through prospective single-center clinical studies, explore the establishment of new predictive models for early diagnosis of severe pneumonia, and optimize the diagnosis and treatment strategy of severe pneumonia, and provide new ideas for accurate treatment of severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥ 18 years, ≤ 75 years, male or female

  * Patients diagnosed with severe pneumonia ③ Immunosuppressed patients

    * Patient informed consent

Exclusion Criteria:

* ① Pregnant women, lactating women and women who are at risk of pregnancy.

  * Patients with malignant neoplasms that have metastasized extensively and are expected to have a short survival period.

    * Patients with obstructive pneumonia and interstitial fibrosis due to lung tumours.

      * refusal of the patient or the patient's family to participate in the study.

        * Refusal of invasive mechanical ventilation and tracheal intubation by the patient or the patient's family.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ICU immunosuppressed pneumonia patients
Sampling Method: Non-Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patient diagnosed with severe pneumonia within 28 days | 28 days